CLINICAL TRIAL: NCT06438991
Title: Epidural Spinal Cord Stimulation for Lower Extremity Motor Function in Spinal Cord Injury
Brief Title: Spinal Cord Stimulation for Lower Extremity Function
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Yi Lu, MD PhD, Director of Neurosurgical Trauma, Associate Professor of Neurosurgery, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2024P000184
Record Dates: First submitted 2024-05-21; First posted 2024-06-03 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Spinal Cord Injury
Keywords: epidural spinal cord stimulation
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: All subjects will receive a spinal cord stimulator. Muscle strength will be assessed with the stimulation turned on and off. Parameters for motor function will be assessed with the stimulation turned on and off.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- All participants (Experimental): Baseline: participants will undergo lower extremity muscle strength testing, electromyography, spine and brain MRI, and complete a battery of questionnaires
  All participants will undergo a clinically indicated spinal cord stimulator implanted for refractory chronic pain.
  SCS Optimization phase consists of weekly research visits for 1 month. SCS parameters will be optimized for voluntary control of lower extremity muscles.
  Individualized Neurorehabilitation phase consists of 4 x weekly visits for 5-months. With the SCS settings turned on for muscle activation, participants will undergo progressive neurorehabilitation by a spinal cord specialized physical therapist.
  All participants who complete the 6-month timepoint will be invited to continue long-term follow up.
  Interventions: Other: Adjustment of spinal cord stimulation parameters for voluntary motor control

INTERVENTIONS:
Other: Adjustment of spinal cord stimulation parameters for voluntary motor control — All patients will receive a spinal cord stimulator and undergo adjustment of stimulation parameters for optimal voluntary lower extremity motor control during research visits. Muscle strength will be assessed with the stimulation turned on and off.

SUMMARY:
This prospective clinical study will investigate the ability of different spine imaging characteristics to predict ambulation recovery responsiveness using epidural spinal cord stimulator (SCS) in patients with chronic incomplete spinal cord injury (SCI).

Epidural spinal cord stimulation below the level of injury can restore previously lost lower extremity voluntary motor function for some patients. The goal of this study is to establish whether spine imaging can be utilized as a biomarker to predict which patients will respond to spinal cord stimulation.

DETAILED DESCRIPTION:
Ten patients with chronic spinal cord injury who are scheduled to receive a spinal cord stimulator for refractory chronic pain will be recruited throughout the Mass General Brigham health system. At baseline, participants will undergo a neurologic strength exam, Magnetic Resonance Imaging (MRI) of the spine and brain, electromyography (EMG) of the lower extremities, and will complete a battery of pain, motor function and quality of life questionnaires.

Phase 1: The SCS Optimization phase consists of weekly research visits during the first month post-SCS implant. Settings of the spinal cord stimulator parameters will be modified for activation and optimal voluntary control of lower extremity muscles.

Phase 2: The Individualized Neurorehabilitation phase consists of 4 weekly visits for a 5-month period. Participants will undergo neurorehabilitation with the stimulation settings turned on for motor control. Neurorehabilitation will be individualized and will progressively increase participants' physical activity, including assisted/independent standing, stepping and ambulation within safe limits. Participants will undergo monthly muscle strength and surface EMG testing.

At the end of each research visit or neurorehabilitation session, SCS settings will be adjusted to the original pain management parameters.

At the 6-month follow up participants will undergo a neurologic strength exam, MRI of the spine and brain, EMG of the lower extremities and a battery of questionnaires. After the last follow up visit, participants will have the opportunity to continue a long-term follow up or exit the study. SCS parameters will be adjusted to the pain management settings.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Provides informed consent
* Eligible for and undergoes SCS implant for chronic low back or leg pain refractory to first-line therapy
* Stable SCI secondary to a single insult
* C6-T10 level of injury
* SCI has occurred >12 months prior to enrollment
* Chronic low back pain refractory to first-line therapy
* Current AIS grade B-C, with spared sensation
* Willingness and ability to adhere to the protocol

Exclusion Criteria:

* History or diagnosis of Central Nervous System malignancy
* Diagnosis that is a contraindication to SCS implantation or surgery
* Diagnosis that precludes the subject from full participation in physical therapy
* Known osteopenia/osteoporosis
* Impairment in post-operative recovery per clinical evaluation by the principal investigator
* Inability to participate in the protocol, including but not limited to all study visits and assessments

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-related adverse events | 0-6 months after baseline
  The primary endpoint of this study is the safety of stimulation parameters for motor function assessed with the number of adverse events for the duration of the study. Relatedness of adverse events to treatment is determined by the principal investigator.

SECONDARY OUTCOMES:
Muscle Strength | 1-6 months after baseline
  The ability to restore previously lost voluntary motor function of the lower extremity will be measured with the Medical Research Council (MRC) grade and compared to baseline. MRC grades range from 0 (no visible muscle contraction) to 5 (normal muscle strength against full resistance). A higher grade indicates a better outcome.
Neuroimaging volumetric measures | 0-6 months after baseline
  Assessment of the functional integrity of corticospinal tracts with spine and brain Magnetic Resonance Imaging (MRI) will be performed at baseline and at the last follow up. MRI volumetric measures are quantified in mm^2.
Voluntary Motor Function | 0-6 months after baseline
  Functional change assessed with the total score on the American Spinal Injury Association Impairment Scale (AIS) of each participant before spinal cord stimulation (SCS) and after SCS augmented with neurorehabilitation therapy. The AIS scale ranges from A (no sensory or motor function is preserved in sacral segments of S4-S5) to E (sensation and motor testing are normal in all segments), with A representing the worst outcome and E representing the best outcome.
Optimized stimulation amplitude for voluntary motor function | 1-6 months after baseline
  Stimulation amplitude required for voluntary motor function measured in mA (miliAmperes) when supine, assisted/independent standing, stepping, walking.
Optimized stimulation frequency for voluntary motor function | 1-6 months after baseline
  Stimulation frequency required for voluntary motor function measured in Hz (Hertz) when supine, assisted/independent standing, stepping, walking.
Optimized stimulation pulse width for voluntary motor function | 1-6 months after baseline
  Stimulation pulse width required for voluntary motor function measured in microseconds when supine, assisted/independent standing, stepping, walking.
Locomotive ability | 1-6 months after baseline
  Ability to stand, step, or walk either assisted or unassisted assessed with the Walking Index for Spinal Cord Injury II (WISCI II) scale. The WISCI II scale ranges from minimum score of 0 (unable to stand) to maximum score of 20 (ambulates with no devices, brace or assistance). A higher score represents a better outcome.
Serious adverse events | 1-6 months after baseline
  Serious adverse events related to the post-SCS implant neurorehabilitation therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Lu, MD, PhD, Study Chair — Brigham and Women's Hospital/Harvard Medical School

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared other than published de-identified data.

REFERENCES:
- [Background] Chalif JI, Chavarro VS, Mensah E, Johnston B, Fields DP, Chalif EJ, Chiang M, Sutton O, Yong R, Trumbower R, Lu Y. Epidural Spinal Cord Stimulation for Spinal Cord Injury in Humans: A Systematic Review. J Clin Med. 2024 Feb 14;13(4):1090. doi: 10.3390/jcm13041090. PMID 38398403
- [Background] Wagner FB, Mignardot JB, Le Goff-Mignardot CG, Demesmaeker R, Komi S, Capogrosso M, Rowald A, Seanez I, Caban M, Pirondini E, Vat M, McCracken LA, Heimgartner R, Fodor I, Watrin A, Seguin P, Paoles E, Van Den Keybus K, Eberle G, Schurch B, Pralong E, Becce F, Prior J, Buse N, Buschman R, Neufeld E, Kuster N, Carda S, von Zitzewitz J, Delattre V, Denison T, Lambert H, Minassian K, Bloch J, Courtine G. Targeted neurotechnology restores walking in humans with spinal cord injury. Nature. 2018 Nov;563(7729):65-71. doi: 10.1038/s41586-018-0649-2. Epub 2018 Oct 31. PMID 30382197
- [Background] Angeli CA, Edgerton VR, Gerasimenko YP, Harkema SJ. Altering spinal cord excitability enables voluntary movements after chronic complete paralysis in humans. Brain. 2014 May;137(Pt 5):1394-409. doi: 10.1093/brain/awu038. Epub 2014 Apr 8. PMID 24713270
- [Background] Calvert JS, Grahn PJ, Strommen JA, Lavrov IA, Beck LA, Gill ML, Linde MB, Brown DA, Van Straaten MG, Veith DD, Lopez C, Sayenko DG, Gerasimenko YP, Edgerton VR, Zhao KD, Lee KH. Electrophysiological Guidance of Epidural Electrode Array Implantation over the Human Lumbosacral Spinal Cord to Enable Motor Function after Chronic Paralysis. J Neurotrauma. 2019 May 1;36(9):1451-1460. doi: 10.1089/neu.2018.5921. Epub 2018 Dec 15. PMID 30430902
- [Background] Darrow D, Balser D, Netoff TI, Krassioukov A, Phillips A, Parr A, Samadani U. Epidural Spinal Cord Stimulation Facilitates Immediate Restoration of Dormant Motor and Autonomic Supraspinal Pathways after Chronic Neurologically Complete Spinal Cord Injury. J Neurotrauma. 2019 Aug 1;36(15):2325-2336. doi: 10.1089/neu.2018.6006. Epub 2019 Mar 6. PMID 30667299